CLINICAL TRIAL: NCT06169852
Title: Stimulus-Evoked Directional Field Potentials to Guide Subthalamic and Pallidal DBS for PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Harrison Walker, MD, Professor of Neurology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300011568; UH3NS130202 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-12-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation; DBS
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: We are investigating unilateral dual-target DBS. The stimulation paradigms utilized include STN DBS alone, GPi DBS alone, and combined STN/GPi DBS.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned each of three different stimulation paradigms for 4 month intervals. Participants and researchers will be blinded to the stimulation paradigm used at any given point in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Arm 1 (0-4 months) (Experimental): In this arm we will stimulate from either STN alone, GPi alone, or a combination of both STN and GPi.
  Interventions: Device: Unilateral dual-target (STN/GPi) DBS
- Arm 2 (4-8 months) (Experimental): In this arm we will stimulate from either STN alone, GPi alone, or a combination of both STN and GPi, whichever was not used in Arm 1.
  Interventions: Device: Unilateral dual-target (STN/GPi) DBS
- Arm 3 (8-12 months) (Experimental): In this arm we will stimulate from either STN alone, GPi alone, or a combination of both STN and GPi, whichever was not used in Arms 1 and 2.
  Interventions: Device: Unilateral dual-target (STN/GPi) DBS

INTERVENTIONS:
Device: Unilateral dual-target (STN/GPi) DBS — Participants will be randomly assigned either DBS stimulation in the STN alone, GPi alone, or a combination of stimulation in the STN and GPi.

SUMMARY:
Our goal is to better understand how DBS modifies local neuronal activity and to pioneer device technologies that can record local DBS-evoked potentials (DLEPs) to guide therapy. Our vision is for a patient's unique electrophysiology to guide both electrode targeting during surgery and programming in clinic, eventually as an integrated component of the implanted pulse generator. Our results will inform directional DBS for PD and serve as a model for translation to other diseases where knowledge on DBS circuit interactions is at an even earlier stage.

DETAILED DESCRIPTION:
This study is an exploratory single center double-blind, randomized crossover study of unilateral STN versus GPi versus dual-target STN/GPi DBS for motor symptoms of PD. The dual-target approach will allow unique measures of connectivity between STN and GPi, and within-participant clinical contrasts of single target STN, single target GPi, and combined dual-target stimulation. Longitudinal encounters will measure changes in motor function, non-motor function, and patient reported outcomes versus pre-operative baseline in response to each of these stimulation conditions at 4-month intervals after surgery. These blinded encounters will be followed by an unblinded open-label encounter at 16 months utilizing optimized stimulation parameters. In addition to the clinical crossover design, we will retrospectively investigate the extent to which the spatial maps of local DBS-evoked potentials within and across brain targets predict stimulation sites chosen for clinical therapy at either brain target.

ELIGIBILITY:
Inclusion criteria:

1. Age >18 years and older.
2. Clinically definite, advanced idiopathic PD based on at least 2 of 3 cardinal PD features (tremor, rigidity, and/or bradykinesia).
3. Disease duration of 4 years or more.
4. Participant has elected to undergo awake DBS surgery as part of routine care, and the subthalamic nucleus (STN) or globus pallidus interna (GPi) are recommended by the multidisciplinary DBS committee as the surgical target.
5. For participants who opt for the dual-target strategy, neurosurgery judges that dual-target STN and GPi implant is an appropriate option with acceptable safety profile.
6. Participant is healthy enough to undergo surgery and the research protocol.
7. Normal, or essentially normal, preoperative brain MRI, except for expected mild abnormalities associated with advanced PD.
8. Willingness and ability to cooperate during awake DBS surgery, as well as during post-operative evaluations, adjustments of medications and stimulator settings.
9. Participant's health insurance and/or Medicare covers DBS surgery as part of routine care.
10. Refractory motor symptoms such as dyskinesias, wearing off, and/or motor fluctuations, causing significant disability or occupational dysfunction, despite reasonable attempts at medical management, as determined by our consensus DBS committee.
11. Stable doses of PD medications for at least 28 days prior to baseline assessments.
12. Improvement of motor signs ≥30% with dopaminergic medication as assessed with the use of the Movement Disorders - Unified Parkinson's Disease Rating Scale, part III (MDS-UPDRS III; scores range from 0 to 108, with higher scores indicating worse functioning). One exception to this 30% threshold is patients who have typical features of PD but cannot take levodopa because of unacceptable side effects.19
13. Disease severity ratings above Hoehn and Yahr stage 2.5, defined as unilateral involvement only with minimal or no functional disability, with scores ranging from 0 to 5 and higher scores indicating more severe disease.
14. Score of more than 6 for activities of daily living in the worst "off" medication condition despite medical treatment, as assessed with the use of the MDS-UPDRS II (scores range from 0 to 52, with higher scores indicating worse functioning), or mild-to-moderate impairment in social and occupational functioning (score of 51 to 80% on the Social and Occupational Functioning Assessment Scale with scores ranging from 1 to 100 and lower scores indicating worse functioning).
15. Dementia Rating Scale-2 (DRS-2) score of ≥130 on medications.
16. Beck Depression Inventory II (BDI-II) score of ≤25 on medications.
17. No indication of suicidal ideation or active suicidal thoughts as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRC).
18. Participant expresses understanding of the consent process, terms of the study protocol, is available for follow-up over the length of the study, and signs informed consent.

Exclusion criteria:

1. Age <18 years.
2. Participant's insurance will not cover the costs of surgery with an investigational device (Aims 2 and 3 only).
3. Medical contraindications such as current uncontrolled hypertension, heart disease, coagulopathy, or other conditions contraindicating DBS surgery or stimulation.
4. Duration of disease of <4 years
5. Clinical team suspects patient will need staged contralateral DBS for clinical symptoms within 1 year of unilateral DBS surgery.
6. Diagnosis or suspicion of atypical parkinsonism (progressive supranuclear palsy, multiple system atrophy, corticobasal syndrome) or drug-induced parkinsonism, or significant neurological disease other than Parkinson's disease.
7. Diagnosis of psychogenic movement disorder based on consensus criteria.
8. Dual-target implant cannot be performed safely from a single burr hole because of anatomic constraints or cortical vascular anatomy, based upon the pre-operative neurosurgery plan.
9. Patient is undergoing DBS electrode placement under general anesthesia without awake electrophysiological and clinical testing during implant.
10. Score of >25 on the Beck Depression Inventory II, with scores ranging from 0 to 63 and higher scores indicating worse functioning), or history of suicide attempt.
11. An indication of suicidal ideation or active suicide planning as assessed on the Columbia-Suicide Severity Rating Scale.
12. Any current acute psychosis, alcohol abuse or drug abuse.
13. Clinical dementia (score of ≤130 on the Mattis Dementia Rating Scale with scores ranging from 0 to 144 and higher scores indicating better functioning).
14. Ongoing or pervasive impulse control disorder not resolved by reduction of dopaminergic medications.
15. Use of anticoagulant medications that cannot be discontinued during perioperative period.
16. History of hemorrhagic stroke.
17. Current or future risk of immunocompromise that might increase infection risk.
18. History of recurrent of unprovoked seizures.
19. Lack of clear levodopa responsiveness.
20. The presence of an implanted device (e.g., cochlear implant, pacemaker, neurostimulators), whether turned on or off.
21. Prior DBS surgery or ablation within the affected basal ganglion.
22. Prior DBS surgery on the opposite side of the brain (Aims 2 and 3 only). This may allow us to study some participants twice (i.e., in Aim 1 or 2-3, and again in Aim 1 if they return for DBS on the opposite side of the brain as part of routine care).
23. A condition requiring or likely to require the use of diathermy.
24. Structural lesions such as basal ganglionic stroke, tumor, or vascular malformation as etiology of the movement disorder.
25. Any medical or psychological problem that would interfere with completing the study protocol, as determined by the research team.
26. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Validate the biological origin of brain signals using an external stimulation/recording system during standard of care Deep Brain Stimulation surgery, both awake and under general anesthesia. | At standard of care DBS surgery (awake) and approximately one week later at standard of care battery placement (under general anesthesia).
  The investigator will validate the biological origin of the signals using pairs of DBS pulses and neural refractoriness with an external stimulation/recording system at therapeutically relevant stimulus amplitudes (i.e., inside and outside the therapeutic window).
Test whether directional DBS leads elicit spatiotemporally distinct oscillations in subthalamic nucleus versus globus pallidus interna. | At standard of care DBS surgery (awake) and approximately one week later at standard of care battery placement (under general anesthesia).
  This investigators efforts will yield granular spatial maps of neural engagement across the two canonical targets for PD to guide targeting (awake or under anesthesia) and clinical programming.
Test whether spatial maps of DBS-evoked oscillations predict clinically effective stimulation sites on a directional DBS lead. | At standard of care DBS surgery (awake), approximately one week later at standard of care battery placement (under general anesthesia), at in a research clinical assessment at 16 months after DBS surgery.
  The investigator will test whether spatial maps of DBS-evoked neural activity predict clinically effective locations for directional DBS.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Walker, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from this project are available upon messaging, email, or written request through the Data Archive for the BRAIN Initiative (PI Dr. Toga at University of Southern California). Coded research data are collected such as electrophysiological signals, clinical rating scales, neuroimaging data, computational analysis algorithms, and biostatistics workflows. The investigator will curate and share these raw data and algorithms via DABI. All data are coded and password-protected to ensure the privacy of human research participants.
Access Criteria: All data resulting from this project are available upon messaging, email, or written request through the Data Archive for the BRAIN Initiative (PI Dr. Toga at University of Southern California).
URL: https://dabi.loni.usc.edu/